CLINICAL TRIAL: NCT00411762
Title: A Phase I/II, Multi-Center, Open-Label, Dose-Escalation, Safety and Efficacy Study of PHY906 Plus Capecitabine in Patients With Advanced Pancreatic Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: PhytoCeutica (Industry); National Comprehensive Cancer Network (Network); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0512000905
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; PHY 906

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PHY906 Administration (Experimental): PHY906 800mg, orally, twice a day for days 1-4 and capecitabine 1500mg/m^2 days 1-7 of a 14-day cycle
  Interventions: Drug: Capecitabine; Drug: PHY906

INTERVENTIONS:
Drug: Capecitabine
  Other Names: Xeloda
Drug: PHY906
  Other Names: Traditional Chinese Medicine: Scutellaria baicalensis Georgi, Glycyrrhiza uralensis Fisch., Ziziphus jujuba Mill., and Paeonia lactiflora Pall

SUMMARY:
The aim of this research project is to determine the amount of capecitabine (Xeloda) which can be given safely with PHY906 (investigational drug) on a novel schedule. It is also the aim of this research project to determine what the effects, good and/or bad, are of combining capecitabine (Xeloda) with PHY906 (investigational drug) in the treatment of advanced pancreatic cancer.

PHY906 is a powder from plants sold as a health food supplement in the United States. PHY906 has been used in China, Taiwan and other Asian countries as traditional Chinese medicine for hundreds of years.

The other drug involved in this study, capecitabine is an oral form of chemotherapy already approved by FDA in the management of colorectal and breast cancer.

Laboratory studies in animal models have shown that the combination of capecitabine and PHY906 shrinks liver cancer, and a pilot clinical study is currently evaluating this combination in patients with liver cancer to define the benefit. PHY906 has also shown to decrease diarrhea related to chemotherapy in a small study performed in patients with colon cancer treated at the Yale Cancer Center. Our recent laboratory studies have also shown that the combination of capecitabine and PHY906 also shrink pancreatic tumors in mouse models. This prompted us to test the combination of capecitabine and PHY906 in patients with advanced pancreatic cancer to assess the benefit in survival as well as any decrease in side effects, such as diarrhea caused by capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years of age with either a histologic or cytologic diagnosis of locally advanced or metastatic pancreatic adenocarcinoma. However, patients with other solid malignancies will be allowed to participate during the dose escalating Phase I part of the study, who had failed to respond to standard therapy or for which no standard therapy exists.
* In the phase I portion, patients may either have had no prior chemotherapy (chemotherapy naive), or have been refractory to or relapsed from standard chemotherapy, including capecitabine-based regimens. However, in the phase II portion of the study, only pancreatic cancer patients with prior gemcitabine therapy will be eligible. No prior 5-FU/capecitabine chemotherapy will be allowed EXCEPT previous adjuvant treatment with 5-FU or capecitabine (radiosensitizing dose) with radiation completed at least 6 weeks prior to study entry.
* All patients in both the phase I and phase II portions of this study must have at least one previously unirradiated, unidimensionally measurable lesion by computerized tomography (CT) or magnetic resonance imaging (MRI) scan of ≥ 20 mm (if conventional CT scan) or ≥ 10 mm (if spiral CT scan).
* Patients with biliary or gastro-duodenal obstruction must have drainage or by pass prior to starting chemotherapy.
* Patients with adequate hepatic function defined as

  * AST/ALT ≤ 2.5 X ULN;
  * Total Bilirubin ≤ 2.0 XULN;
  * Alkaline Phosphatase ≤ 5 X ULN (in presence of liver metastasis); or
  * Alkaline Phosphatase ≤ 2.5 X ULN (in absence of liver metastasis).
* Patients should have an adequate renal function as indicated by a serum creatinine <1.6 mg/dL or calculated creatinine clearance ≥ 50 mL/min. (Calculated by Cockcroft-Gault equation).
* Baseline performance status must be Eastern Cooperative Oncology Group (ECOG) 0, 1, or 2.
* Women patients who are known to be capable of conception should have a negative serum pregnancy test (beta-human chorionic gonadotropin [beta-hCG]) within 2 weeks of starting the study; all patients should agree to use adequate non-estrogenic birth control methods, consistent with the institute's standard form of contraception if conception is possible during the study.
* Provide written informed consent prior to screening.
* Patients with adequate hematologic tests:

  * Hemoglobin ≥ 9.0 g/dL;
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10 9/L;
  * Platelet count ≥ 100.0 x 10 9/L;

Exclusion Criteria:

* Patients who are pregnant or breastfeeding.
* Any prior palliative radiation therapy (other than used in the adjuvant therapy of pancreatic cancer > 6 weeks) must have been completed more than 21 days before entry into the study and evaluable lesions must not have been included in the radiation portal.
* Patients with prior capecitabine therapy for pancreatic cancer (Phase II).
* Patients with active CNS metastases.
* Patients with known hypersensitivity or a history of marked intolerance to 5-FU are ineligible.
* Because cimetidine can decrease the clearance of 5-FU, patients should not enter on this study until cimetidine is discontinued.
* Patients should not receive concurrent therapy with either sorivudine or brivudine, while receiving capecitabine. If a patient has received prior sorivudine or brivudine, then at least four weeks must elapse before the patient receives capecitabine therapy.
* Exclude sexually active males unwilling to practice contraception during the study.
* Lack of physical integrity of the upper gastrointestinal tract, inability to swallow tablets or those who have malabsorption syndrome.
* Clinically significant cardiac disease not well controlled with medication (e.g., congestive heart failure, symptomatic coronary artery disease, and cardiac arrhythmias) or myocardial infarction within the last 12 months.
* No concurrent radiotherapy is allowed.
* Known DPD (dihydropyrimidine dehydrogenase) deficiency.
* Patients who have received any previous treatment consisting of standard chemotherapy (gemcitabine in Phase II study; others in Phase I) within 21 days or an investigational agent (Phase I) within 30 days on study. Toxicity related to the previous therapy must have resolved prior to study entry.
* Patients with previous or concurrent malignancy except for inactive non-melanoma skin cancer and/or in situ carcinoma of the cervix, or other solid tumor treated curatively and without evidence of recurrence within the last 3 years prior to study entry.
* Patients taking herbal medicine(s), including supplement(s), are eligible if they discontinue the herbal medicine(s)/supplement(s) at least 7 days prior to study entry.
* Known allergy or hypersensitivity to PHY906 or any of the components used in the PHY906 formulations, or to capecitabine.
* Serious concurrent medical illness, which would jeopardize the ability of the patient to receive the chemotherapy program outlined in this protocol with reasonable safety.
* Patients with active infections requiring intravenous antibiotic therapy are not eligible until the infection has resolved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Hochester, MD, Principal Investigator — Yale University
Locations (1):
- Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PHY906 Administration: PHY906 800mg, orally, twice a day for days 1-4 and capecitabine 1500mg/m^2 days 1-7 of a 14-day cycle
  Capecitabine
  PHY906
Period: Overall Study
Arm/Group | PHY906 Administration
Started | 25
Completed | 20
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | PHY906 Administration
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 64 [45 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 100 weeks
Population: 20 subjects received 2 cycles or more and were evaluated for response
Measure: Median (Full Range); unit: weeks
Groups:
- PHY906 Administration: PHY906 800mg, twice a day for days 1-4 and capecitabine 1500mg/m^2 days 1-7 of a 14-day cycle
Arm/Group | PHY906 Administration
Number analyzed (Participants) | 20
weeks | 10.1 [0.4 to 54.1]

2. Secondary Outcome: Median Overall Survival
Description: as for outcome 1
Time Frame: Up to 100 weeks
Population: 20 subjects received 2 cycles or more and were evaluated for response
Measure: Median (Full Range); unit: weeks
Arm/Group | PHY906 Administration
Number analyzed (Participants) | 20
weeks | 21.6 [0.4 to 84.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the duration of the study (approximately 4 years)
Arm/Group | PHY906 Administration
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 10/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PHY906 Administration (N=25)
Anemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Mucositis (Skin and subcutaneous tissue disorders) | 4
Anorexia (Gastrointestinal disorders) | 8
Dry mouth/taste alternation (General disorders) | 2
Nausea/vomiting (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 7
Hand-Foot Syndrome (General disorders) | 5
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Elevated Liver Function Tests (Hepatobiliary disorders) | 2
Electrolytes Imblances (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes